CLINICAL TRIAL: NCT03520933
Title: A Prospective, Observational, Multi-center, International Study to Validate a Non-invasive Preimplantation Genetic Test for Embryo Aneuploidy in the Spent Culture Media (niPGT-A).
Brief Title: Multi-center Study to Validate niPGT-A
Acronym: niPGT-A
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-NIP-CS-18-02-SUB1
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Aneuploidy; Chromosome Abnormality; Infertility
Keywords: Embryo; Blastocyst; Non-invasive; PGT-A; Chromosome; Aneuploidy; Spent culture medium; Trophectoderm biopsy
MeSH Terms: conditions — Aneuploidy; Chromosome Aberrations; Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Culture media: Embryonic cell-free DNA (cfDNA)
  * Trophectoderm biopsy
  * Inner cell mass biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Embryos undergoing PGT-A / niPGT-A: Embryos from IVF patients between 20 and 44 years of age, undergoing PGT-A for any medical indication, with own oocytes or ovum donation cycles and with single embryo transfer (SET)
  Interventions: Diagnostic Test: PGT-A; Diagnostic Test: niPGT-A

INTERVENTIONS:
Diagnostic Test: PGT-A — PGT-A will be carried out following the usual clinical practice: Trophectoderm biopsy samples from blastocysts are analyzed by NGS to screen for numerical chromosomal abnormalities.
Diagnostic Test: niPGT-A — Non-invasive preimplantation genetic test for embryo aneuploidy analyzing the spent culture media where the embryo is incubated up to the time of vitrification. This media contains traces of embryonic cell-free DNA (cfDNA) that can represent the genetic load of the embryo.

SUMMARY:
Abnormal chromosome number, or aneuploidy, is common in human embryos. It is responsible for more than half of all miscarriages, and it is the leading cause of congenital birth defects. Besides, it has been described that aneuploidy may also affect embryo implantation. Therefore, selecting embryos that have the best chance of implanting and growing into a healthy baby is one of the most important steps in the field of assisted reproduction.

Recent advances in genetic technologies, such as Next-Generation Sequencing (NGS), have allowed aneuploidy to be detected with greater sensitivity. The application of this technique to trophectoderm biopsies, taken from embryos before transfer to the uterus, has provided insight into the clinical impact of chromosomal status. This process of screening embryos to make sure they have the right number of chromosomes and to look for any structural abnormalities in the chromosomes is called Preimplantation Genetic Testing for Aneuploidy (PGT-A). It requires specific equipment and trained personnel that will add costs and risks, so non-invasive techniques are sought as an alternative. These non-invasive procedures have been explored by some groups analyzing the spent culture medium where the embryo is cultured up to the time of transfer or freezing. In daily routine, this media is discarded after finishing the embryo culture, but it has been reported that contains traces of embryonic cell-free DNA (cfDNA) that can represent the genetic load of the embryo. However, at the moment there is a high variability in results across studies, with a percentage of concordant results between the media and the trophectoderm biopsy ranging from 3.5 to 85.7%.

Thus, the main objective of this project is to validate a new non-invasive method for PGT-A (niPGT-A), based on improved collection and analysis of the culture media to achieve higher rates of sensitivity and specificity and to decrease the effect of some intrinsic difficulties such as low embryonic cfDNA input, mosaicism and maternal contamination.

DETAILED DESCRIPTION:
Human embryos have higher aneuploidy rates (20-80%) than other species. A considerable proportion of these aneuploid embryos have the ability to reach the blastocyst stage. However, depending on the aneuploidy type, some will fail to implant in the uterus, while others will implant but will be unable to carry out early embryonic development (miscarriage), or very rarely, result in liveborn children with specific abnormalities. It is therefore important to identify aneuploid embryos. The identification of aneuploidies is especially important in embryos from patients with higher aneuploidy risk such as those with advanced maternal age (AMA), recurrent implantation failure (RIF), or recurrent miscarriage (RM).

PGT-A technique analyse the full chromosome content of the embryo with high sensitivity and specificity but requires an invasive biopsy to obtain embryonic material for the genetic analysis. Thus, non-invasive methods to replace the existing invasive testing method would be useful in the improvement of maternal and fetal safety.

Recently, there have been many research advances in the field of genetic testing. Cell-free DNA (cfDNA) has been observed in spent embryo culture media. The origin of the cfDNA at the blastocyst stage remains unknown and this has encouraged different research groups to carry out analysis of the spent culture media.

Various studies were initially carried out to detect specific genes associated with monogenic disorders (MTHFR9, HBA1/HBA210, SRY11). Recently, non-invasive PGT-A has been developed, with highly variable results on the concordance rate (3.5%,59.1%, and 85.7%, 30.6%). The chromosomal status of the embryo from the DNA present in the spent culture medium was compared to the one obtained following the standard protocol using trophectoderm biopsy. The difference in the reported results can be related to the different methodologies applied because different amplification and detection methods -aCGH or NGS- were used. Moreover, the concordance rates were defined differently on each study, i.e. aneuploid results in spent culture media and trophectoderm biopsy could be considered concordant despite of showing not the same aneuploid chromosomes.

The impact of culture conditions in the efficiency of the non-invasive approach has been thoroughly investigated. There could be influence of these relevant factors: external contamination from laboratory personnel or equipment, contamination with maternal DNA from granulosa cells (MCC) and mosaicism threshold for diagnosis..

To improve the results of IVF (In vitro Fertilization) programs, there is a need to identify the embryo with highest implantation potential. Embryo chromosomal analysis allows the selection of euploid embryos, which have a higher implantation success rate.

The development of a non-invasive PGT-A protocol will improve the current methodologies used to identify those euploid embryos avoiding the detrimental effect of the biopsy on the embryo and decreasing the economic cost.

The main objective of the current study is to validate a new non-invasive method for PGT-A (niPGT-A), based on improved collection and analysis of the culture media to achieve higher rates of sensitivity and specificity and to decrease the effect of some intrinsic difficulties such as low embryonic cfDNA input and maternal contamination. The initial estimated sample size calculated was 3245embryos (each embryo is considered as a subject in the study), considering a dropout rate of 30%.

Data exported from the medical records and source documents will be duly codified to protect the clinical and personal information of patients in accordance with the current legislation. This information will be exported to an electronic Case Report Form (eCRF). Data will be grouped and analyzed at Igenomix at three time points of the study: once 25 embryos of each center have been processed (to assess the implementation of the methodology), after the 30% of the samples have been processed (as an interim to check the results) and at the end of the study for the final analysis including the follow up of the clinical outcomes (defined following The International Glossary on Infertility and Fertility Care, 2017).

After the interim analysis, the total sample size has been recalculated as 2620 samples, considering a drop-out rate of 5% according to the drop-out rate observed. Results of the interim analysis were published in Rubio et al., AJOG 2020.

ELIGIBILITY:
Inclusion Criteria:

* PGT-A cases with trophectoderm biopsy and SET for any medical indication and signed written informed consent form approved by the EC/IRB after having been duly informed of the nature of the research and voluntarily accepted to participate in the study.
* ICSI (Intra Cytoplasmic Sperm Injection), IVF (In Vitro Fertilization) or ICSI/IVF performed in fresh oocytes from couples are allowed.

Note: Donor sperm is allowed.

* Only fresh oocytes allowed.
* Fresh and Deferred Embryo Transfer are allowed. Note: In case of Deferred Embryo Transfer, embryos must be vitrified always after the blastocyst biopsy.
* Age: 20-44 years of age (both included).

Exclusion Criteria:

* A known abnormal karyotype in a member of the couple.
* Preimplantation Genetic Testing for Monogenic diseases (PGT-M) or Preimplantation Genetic Testing for Structural Rearrangements (PGT-SR) cases excluded.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — IVF patients
Study Population: Embryos from IVF patients between 20 and 44 years of age, undergoing PGT-A for any medical indication, with own oocytes or ovum donation cycles and with single embryo transfer (SET).
Sampling Method: Non-Probability Sample
Enrollment: 2586 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Chromosomal status of the embryos | 6 to 7 days of embryo development
  Concordance on number and structure of the chromosomes between biopsy and spent blastocyst media samples analysis results.

SECONDARY OUTCOMES:
Pregnancy rate | 20 weeks
  Number of pregnancies per embryo transfer
Clinical miscarriage rate | 20 weeks
  Number of clinical miscarriages per total number of pregnancies
Analysis of the Products of Conception (POC) | Up to 20 weeks
  Placental and/or fetal tissue that remains in the uterus after a spontaneous pregnancy loss
Live birth rate | 40 weeks
  Number of babies born per embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Rubio, BSc PhD, Principal Investigator — Igenomix; Carlos Simón, MD PhD, Study Chair — Igenomix
Locations (10):
- United States (3):
  - San Diego Fertility Center, San Diego, California
  - Boston IVF Fertility Clinic, Boston, Massachusetts
  - Dominion Fertility, Arlington, Washington
- Pregna Medicina Reproductiva, Buenos Aires, Argentina
- Nilo Frantz - Centro de Reprodução Humana, Boa Vista, Porto Alegre, Brazil
- Genera Rome, Rome, Roma, Italy
- NASCERE, Mexico City, Mexico City, Mexico
- Inmater - Clínica de Fertilidad, Lima, Peru
- ProcreaTec, Madrid, Spain
- Bahçeci Group, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakkas D, Navarro-Sanchez L, Ardestani G, Barroso G, Bisioli C, Boynukalin K, Cimadomo D, Frantz N, Kopcow L, Andrade GM, Ozturk B, Rienzi L, Weiser A, Valbuena D, Simon C, Rubio C. The impact of implementing a non-invasive preimplantation genetic testing for aneuploidies (niPGT-A) embryo culture protocol on embryo viability and clinical outcomes. Hum Reprod. 2024 Sep 1;39(9):1952-1959. doi: 10.1093/humrep/deae156. PMID 39059790